CLINICAL TRIAL: NCT07161492
Title: Effects of Repetitive Transcranial Magnetic Stimulation (rTMS) on Cognitive Flexibility and Brain Functional Connectivity in Patients With Major Depressive Disorder: A Randomized Controlled Trial
Brief Title: A Study on Functional Connectome and rTMS Intervention of Cognitive Flexibility Impairment in Patients With Major Depressive Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KYZ20250118
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Depressive Disorder, Major; Cognitive Impairment
MeSH Terms: conditions — Depressive Disorder, Major; Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation; Selective Serotonin Reuptake Inhibitors; Serotonin and Noradrenaline Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CCRT+TAU (Experimental): Participants receive:
  1. Computerized Cognitive Remediation Therapy (CCRT):
     * Cognitive flexibility module (4-6 exercises per session)
     * 45-60 min/session, 5 sessions/week for 4 weeks
     * Difficulty progression based on performance
  2. Treatment As Usual (TAU):
     * Stable-dose SSRIs/SNRIs (e.g., paroxetine 20-40mg/day)
     * Continued throughout study"
  Interventions: Behavioral: Computerized Cognitive Remediation Therapy; Drug: Selective Serotonin Reuptake Inhibitors or Serotonin-Norepinephrine Reuptake Inhibitors
- TAU Control (Active Comparator): Participants receive:
  * Treatment As Usual (TAU) only:
  * Stable-dose SSRIs/SNRIs (e.g., paroxetine 20-40mg/day)
  * No CCRT intervention"
  Interventions: Drug: Selective Serotonin Reuptake Inhibitors or Serotonin-Norepinephrine Reuptake Inhibitors
- Active rTMS+TAU (Experimental): Participants receive:
  1. Individualized dual-target rTMS:
     * Target: Left IPL-right dPFC connectivity (fMRI-guided)
     * Protocol: cc-PAS (100 pulse-pairs/session, 0.2Hz)
     * Intensity: 90-120% resting motor threshold
     * Duration: 8.3 min/session, 5 sessions/week for 4 weeks
     * Device: MagPro X100 with Cool-B65 coil
  2. Treatment As Usual (TAU):
     * Stable-dose SSRIs/SNRIs"
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Drug: Selective Serotonin Reuptake Inhibitors or Serotonin-Norepinephrine Reuptake Inhibitors
- Sham rTMS+TAU (Sham Comparator): Participants receive:
  1. Sham rTMS:
     * Identical setup as active arm
     * Coil tilted 90° with magnetic shield
     * Sound/sensation matched
  2. Treatment As Usual (TAU):
     * Stable-dose SSRIs/SNRIs"
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation; Drug: Selective Serotonin Reuptake Inhibitors or Serotonin-Norepinephrine Reuptake Inhibitors

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Individualized dual-target rTMS delivered using MRI-guided neuronavigation (Dolphin Robotics). Stimulation parameters:
  * Targets: Left IPL and right dPFC connectivity hotspots
  * Protocol: 100 pulse-pairs/session at 0.2Hz
  * Intensities: Conditioning stimulus 90% RMT, test stimulus 120% RMT
  * Duration: 8.3 min/session, 5 sessions/week × 4 weeks
  Arms: Active rTMS+TAU
Behavioral: Computerized Cognitive Remediation Therapy — Structured computer-based training targeting cognitive flexibility, consisting of 4-6 exercises per session. Each exercise includes 8-24 progressively challenging tasks. Administered for 45-60 minutes per session, 5 sessions/week over 4 weeks. Delivered via specialized software on desktop computers.
  Arms: CCRT+TAU
Device: Sham Repetitive Transcranial Magnetic Stimulation — Inactive stimulation using identical equipment with:
  * Coil tilted at 90° to scalp
  * Magnetic shielding insert
  * Matched acoustic artifact All other parameters identical to active rTMS arm.
  Arms: Sham rTMS+TAU
Drug: Selective Serotonin Reuptake Inhibitors or Serotonin-Norepinephrine Reuptake Inhibitors — Background antidepressant therapy maintained at stable doses throughout the study. Minimum dose requirements:
  * SSRIs: Paroxetine ≥20mg/day, Sertraline ≥50mg/day
  * SNRIs: Venlafaxine ≥75mg/day, Duloxetine ≥60mg/day Dosage adjustments prohibited during trial participation.

SUMMARY:
Persistent cognitive impairment in major depressive disorder (MDD) affects both treatment outcomes and psychosocial functioning, emphasizing the critical need for effective treatment. However, there is still a lack of effective treatment at present. Our previous studies found that the impairment in cognitive flexibility (CF) persisted even in remitted patients with MDD. This impairment was correlated with hypo-connectivity between the left inferior parietal lobule (IPL) and the right dorsal prefrontal cortex (dPFC). Based on these findings, we hypothesize that the hypo-connectivity between the left IPL and the right dPFC is the neural basis of CF impairment, and targeted interventions of this connection may alleviate CF impairment and thus improve treatment outcomes as well as psychosocial functioning of patients with MDD. The present study proposes to employ cognitive training for MDD patients with CF impairment. By comparing changes in CF and brain functional connectivity via task-based fMRI before and after the intervention, we aim to clarify the effect of cognitive training on cognitive performance, treatment outcomes and psychosocial functioning, and identify the critical role of the hypo-connectivity between the left IPL and the right dPFC underlying CF impairment. Furthermore, we will conduct a randomized controlled trial to investigate the effect of individualized dual-target repetitive transcranial magnetic stimulation (rTMS) on CF by targeting the hypo connectivity between the left IPL and the right dPFC. The results will further validate the critical role of this connection in modulating CF performance and provide a reliable intervention target for reducing CF impairment.

DETAILED DESCRIPTION:
This is a mechanistic clinical trial investigating the neural basis of cognitive flexibility (CF) impairment in major depressive disorder (MDD) and the therapeutic effects of targeted neuromodulation. The study consists of three integrated components:

1. Component 1 (RCT: CCRT vs. TAU)

   MDD patients with CF impairment will be randomized to:
   * Arm A: Computerized Cognitive Remediation Therapy (CCRT) targeting CF + Treatment As Usual (TAU)
   * Arm B: TAU alone Objective : Examine whether CCRT improves CF and whether CF improvement translates to better clinical/functional outcomes.
2. Component 2 (Neuroimaging Biomarker Study)

   Cross-sectional comparison of:
   * CF-impaired MDD patients
   * CF-intact MDD patients Objective : Identify functional connectivity (FC) signatures of CF impairment using task-based fMRI during cognitive flexibility tasks.
3. Component 3 (RCT: Active vs. Sham rTMS)

CF-impaired MDD patients will be randomized to:

* Arm C: Individualized dual-target rTMS (left IPL-right dPFC) + TAU
* Arm D: Sham rTMS + TAU Objective : Test whether cc-PAS rTMS normalizes left IPL-right dPFC hypo-connectivity and improves CF.

Scientific Rationale :

Hypo-connectivity between left inferior parietal lobule (IPL) and right dorsal prefrontal cortex (dPFC) is hypothesized to be a key neural mechanism underlying persistent CF impairment in MDD. This study aims to:

* Validate this circuit as a therapeutic target
* Establish fMRI-guided cc-PAS rTMS as a precision intervention

Methodology :

Individualized targeting : fMRI-guided neuronavigation (Dolphin Robotics) to identify subject-specific IPL/dPFC coordinates Novel stimulation : Cortico-cortical paired associative stimulation (cc-PAS) to modulate directional connectivity Cognitive phenotyping : Wisconsin Card Sorting Test (WCST) and Trail Making Test (TMT-B/A) as primary CF measures

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-5 criteria for Major Depressive Episode confirmed by two attending psychiatrists using SCID-5
2. Currently in depressive episode (MADRS ≥22)
3. Stable dose of SSRIs/SNRIs for ≥4 weeks prior to randomization
4. Age 18-45 years
5. Han Chinese ethnicity, right-handed
6. Minimum junior high school education; no color blindness; capable of providing informed consent
7. Willing to sign informed consent and complete all assessments

Exclusion Criteria:

1. Other DSM-5 psychiatric disorders (except MDD)
2. Received non-pharmacotherapy in past 6 months:

   * ECT
   * rTMS
   * Systematic psychotherapy (>10 sessions)
3. Prior CCRT treatment
4. Medications affecting cognition within specified washout periods:

   * Antipsychotics (1 month)
   * Cholinesterase inhibitors (donepezil:14d; galantamine:2d)
   * Memantine (20d)
   * Nootropics (e.g., piracetam:2d)
5. Significant medical comorbidities:

   * Thyroid disorders, SLE, diabetes
   * Hepatic/renal/pulmonary impairment
   * Active infections
   * Major trauma
6. History of traumatic brain injury with coma
7. Substance/alcohol abuse or dependence
8. Active suicidal ideation/attempt (MADRS item 10 ≥4)
9. Current corticosteroid therapy
10. Pregnancy, lactation, or planned pregnancy
11. Personal/family history of epilepsy
12. Metallic implants (e.g., pacemaker, dental prostheses)
13. Investigator-determined contraindications

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 182 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive flexibility assessed by Trail Making Test Part B minus Part A (TMT B-A) | Baseline to 4 weeks
  Time difference in seconds between completion of TMT-B and TMT-A. Higher values indicate greater impairment in cognitive flexibility. Measured at baseline and 4 weeks post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Second Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen Y, Liu J, Li Z, Liu B, Ji Y, Ju Y, Fang H, Zheng Q, Wang M, Guo W, Li H, Lu X, Li L. The Tendency of Modified Electroconvulsive Therapy-Related Working Memory and Subjective Memory Deficits in Depression: A Prospective Follow-up Study. J ECT. 2020 Sep;36(3):198-204. doi: 10.1097/YCT.0000000000000668. PMID 32118689
- [Background] Liu J, Dong Q, Lu X, Sun J, Zhang L, Wang M, Liu B, Ju Y, Wan P, Guo H, Zhao F, Zhang X, Zhang Y, Li L. Influence of comorbid anxiety symptoms on cognitive deficits in patients with major depressive disorder. J Affect Disord. 2020 Jan 1;260:91-96. doi: 10.1016/j.jad.2019.08.091. Epub 2019 Aug 29. PMID 31493645
- [Background] Ju Y, Horien C, Chen W, Guo W, Lu X, Sun J, Dong Q, Liu B, Liu J, Yan D, Wang M, Zhang L, Guo H, Zhao F, Zhang Y, Shen X, Constable RT, Li L. Connectome-based models can predict early symptom improvement in major depressive disorder. J Affect Disord. 2020 Aug 1;273:442-452. doi: 10.1016/j.jad.2020.04.028. Epub 2020 May 11. PMID 32560939
- [Background] Wang M, Ju Y, Lu X, Sun J, Dong Q, Liu J, Zhang L, Zhang Y, Zhang S, Wang Z, Liu B, Li L. Longitudinal changes of amplitude of low-frequency fluctuations in MDD patients: A 6-month follow-up resting-state functional magnetic resonance imaging study. J Affect Disord. 2020 Nov 1;276:411-417. doi: 10.1016/j.jad.2020.07.067. Epub 2020 Jul 20. PMID 32871671
- [Background] Liu J, Fan Y, Ling-Li Zeng, Liu B, Ju Y, Wang M, Dong Q, Lu X, Sun J, Zhang L, Guo H, Futao Zhao, Weihui Li, Zhang L, Li Z, Liao M, Zhang Y, Hu D, Li L. The neuroprogressive nature of major depressive disorder: evidence from an intrinsic connectome analysis. Transl Psychiatry. 2021 Feb 4;11(1):102. doi: 10.1038/s41398-021-01227-8. PMID 33542206
- [Background] Liu J, Ju Y, Fan Y, Liu B, Zeng LL, Wang M, Dong Q, Lu X, Sun J, Zhang L, Guo H, Zhao F, Li W, Zhang L, Li Z, Liao M, Zhang X, Zhang Y, Hu D, Li L. Functional connectivity evidence for state-independent executive function deficits in patients with major depressive disorder. J Affect Disord. 2021 Aug 1;291:76-82. doi: 10.1016/j.jad.2021.04.080. Epub 2021 May 21. PMID 34023750
- [Background] Guo W, Liu J, Liu B, Wang M, Dong Q, Lu X, Sun J, Zhang L, Guo H, Zhao F, Li W, Li Z, Liao M, Zhang L, Zhang Y, Ju Y, Li L. Relationship between childhood maltreatment and cognitive function in medication-free patients with major depressive disorder. Eur Arch Psychiatry Clin Neurosci. 2023 Aug;273(5):1073-1083. doi: 10.1007/s00406-022-01458-w. Epub 2022 Jul 29. PMID 35902412
- [Background] Ju Y, Wang M, Liu J, Liu B, Yan D, Lu X, Sun J, Dong Q, Zhang L, Guo H, Zhao F, Liao M, Zhang L, Zhang Y, Li L. Modulation of resting-state functional connectivity in default mode network is associated with the long-term treatment outcome in major depressive disorder. Psychol Med. 2023 Oct;53(13):5963-5975. doi: 10.1017/S0033291722002628. Epub 2022 Sep 27. PMID 36164996
- [Background] Liu J, Chen Y, Xie X, Liu B, Ju Y, Wang M, Dong Q, Lu X, Sun J, Zhang L, Guo H, Zhao F, Li W, Zhang L, Li Z, Liao M, Li L, Zhang Y. The percentage of cognitive impairment in patients with major depressive disorder over the course of the depression: A longitudinal study. J Affect Disord. 2023 May 15;329:511-518. doi: 10.1016/j.jad.2023.02.133. Epub 2023 Feb 28. PMID 36863474
- [Background] Liu J, Zhao X, Wei X, Yan D, Ou W, Liao M, Ji S, Peng Y, Wu S, Wang M, Ju Y, Zhang L, Li Z, Liu B, Li L, Zhang Y. Empirical evidence for the neurocognitive effect of nitrous oxide as an adjunctive therapy in patients with treatment resistant depression: A randomized controlled study. Psychiatry Res. 2023 Aug;326:115326. doi: 10.1016/j.psychres.2023.115326. Epub 2023 Jun 26. PMID 37390601
- [Background] Guo W, Liu B, Wei X, Ju Y, Wang M, Dong Q, Lu X, Sun J, Zhang L, Guo H, Zhao F, Li W, Li Z, Liao M, Zhang L, Liu J, Zhang Y, Li L. The longitudinal change pattern of cognitive subtypes in medication-free patients with major depressive disorder: a cluster analysis. Psychiatry Res. 2023 Sep;327:115413. doi: 10.1016/j.psychres.2023.115413. Epub 2023 Aug 12. PMID 37579539